CLINICAL TRIAL: NCT01438970
Title: Effects of Treatment of Ascites by the ALFApump System on Renal and Circulatory Function in Patients With Cirrhosis and Recurrent or Refractory Ascites
Brief Title: Effects of Treatment of Ascites by the ALFApump System on Renal and Circulatory Function
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-AAR-003
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Cirrhosis, Liver; Refractory Ascites
MeSH Terms: conditions — Liver Cirrhosis; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALFApump system implantation (Other): Implantation of ALFApump system
  Interventions: Device: ALFApump system

INTERVENTIONS:
Device: ALFApump system — The device described above will be implanted using general anaesthesia. The device will be programmed according to each patient's individual requirements, setting the daily loss of ascitic fluid needed to maintain a stable body weight.

SUMMARY:
This is a single centre, prospective, uncontrolled study to include 12 consecutive patients with cirrhosis of the liver and recurrent or refractory ascites. The main aim (primary objective) of the study is to investigate the effect of treatment of ascites by the Sequana medical pump on the renal and circulatory function in patients with cirrhosis and recurrent or refractory ascites. The secondary objectives are the following:

* To evaluate the efficacy of treatment for handling ascites, associated with changes in the body weight of patients and their requirements for evacuation paracentesis during follow-up.
* To investigate the effects of treatment on bacterial translocation, by means of determining bacterial DNA.
* To determine the incidence of complications associated with treatment in the course of follow-up.
* To evaluate the effect of treatment on quality of life of the patients treated, evaluated in questionnaires entitled Short Form-36 and CLDQ (chronic liver disease questionnaire).

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age
2. Cirrhosis of the liver defined by histological and/or clinical, analytical and radiological criteria.
3. Presenting refractory or recurrent ascites, requiring 2 or more evacuation paracentesis procedures over the last 3 months.
4. Written informed consent
5. Ability to comply with study procedures and ability to operate the device
6. Women of childbearing age should use adequate contraceptives

Exclusion Criteria:

1. Digestive haemorrhage over the last 7 days (these patients can be included once the 7-day period has gone by).
2. Kidney failure defined as serum creatinine higher than or equal to 2 mg/dl.
3. Serum bilirubin greater than 5 mg/dl.
4. Severe coagulopathy defined as platelet count of less than 40,000 or prothrombin time of less than 40%.
5. Recurring bacterial peritonitis, defined as 2 or more episodes over the last 6 months.
6. Recurring urinary infections, defined as 2 or more episodes over the last 6 months.
7. Clinical evidence of loculated ascites.
8. Advanced hepatocarcinoma, defined as one which exceeds Milan criteria.
9. Previous liver transplant.
10. Obstructive uropathy or any bladder anomaly which might contraindicate implantation of the device.
11. Pregnancy
12. Patients being in another clinical study that did not reach primary endpoint yet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The main aim of the study is to investigate the effect of treatment of ascites by the Sequana medical pump on the renal and circulatory function in patients with cirrhosis and recurrent or refractory ascites. | One month

CONTACTS AND LOCATIONS:
Overall Officials: Pere Gines, MD, Principal Investigator — Hospital Clinica Barcelona, Spain
Locations (1):
- Hospital clinic, Barcelona, Spain